CLINICAL TRIAL: NCT00939523
Title: Targeted Therapy With Lapatinib in Patients With Recurrent Pituitary Tumors Resistant to Standard Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Odelia Cooper, Principal investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18129
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pituitary Adenomas; Prolactinomas
Keywords: recurrent nonfunctioning adenoma; prolactinomas; resistant pituitary tumors; aggressive pituitary tumors; malignant pituitary adenomas
MeSH Terms: conditions — Pituitary Neoplasms; Prolactinoma | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lapatinib (Experimental): All participants will be asked to take Lapatinib daily for a total of six months during the research study.
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — All participants will be asked to take Lapatinib daily for six months during the research study.
  Other Names: Tykerb

SUMMARY:
This study focuses on new therapies for a challenging disease in pituitary medicine, that of aggressive pituitary tumors which have limited therapeutic options beyond standard surgical, radiotherapy, and select medical therapies, each incurring significant morbidity and mortality, and each not optimally effective. To improve this gap in knowledge, we seek to translate findings from the laboratory into clinical practice and hone in on therapies directed at pituitary molecular targets, namely ErbB receptors. We have shown that human prolactinomas express nuclear EGFR and membranous ErbB2, ErbB3 and ErbB4, and expression correlates with tumor invasion. Pituitary tumor cell lines transfected with EGFR and ErbB2 translated to downstream effects on prolactin (PRL) gene expression and secretion,as well as cell proliferation. Animal models implanted with these cell lines developed larger tumors and PRL elevations. Treatment with ErbB tyrosine kinase inhibitors (TKIs) led to regression of tumors xenografted into these animals and attenuated PRL secretion. Primary culture of human prolactinomas confirmed expression of ErbB receptors and inhibitory effects of TKIs on PRL secretion and cell proliferation. Based on these exciting preliminary data, the objective of this new proposal is to conduct a Phase IIa clinical trial as a trenchant test of our translational hypothesis that tyrosine kinase inhibition constitutes highly effective targeted biologic therapy for these hitherto refractory pituitary adenomas. Specifically, our aims are to test the: 1) efficacy of TKI therapy with a clinical trial; 2) threshold level of tumor receptor expression to achieve TKI clinical response. Nineteen subjects will be treated with lapatinib for 6 months in combination with their current dopamine agonist therapy, with monthly measurements of PRL levels and MRI imaging every 3 months to evaluate the primary endpoints of achieving 40% reduction in tumor size and 50% reduction in PRL and secondary endpoints of radiologic stabilization and/or reduction and PRL normalization. Mean ErbB receptor protein expression will be compared between responders to lapatinib and non-responders by immunohistochemistry in pituitary tumor samples of these subjects collected from prior surgeries.

DETAILED DESCRIPTION:
PURPOSE

The drug Lapatinib has been shown to inhibit both epidermal growth factor receptor (EGFR) and erbB2 tyrosine kinases resulting in an effective slowing of disease progression in breast cancer. It has also been demonstrated that erbB is overexpressed in human pituitary adenomas. The investigators are therefore assessing tumor size stabilization and pituitary tumor secretory profiles during the course of a six month therapy of lapatinib. The purpose of this trial will be to estimate the activity of lapatinib in slowing the growth rate of pituitary tumors. Lapatinib is an FDA approved drug used to treat breast cancer. However, in this study, the drug will be used to treat pituitary cancer.

STUDY POPULATION

This study will recruit patients from the Pituitary Center at CSMC who are over the age of 18 that have a recurrent nonfunctioning adenoma after at least one surgical resection as well as patients with prolactinomas who are resistant to dopamine agonist therapy and patients with recurrent Cushing's disease.

PARTICIPANT'S JOURNEY THROUGH THE RESEARCH

The principal investigator (PI) or co-investigator will determine patients' potential eligibility for the study based on inclusion and exclusion criteria.

The PI or the co-investigator will then approach subjects with recurrent nonfunctioning adenomas or prolactinomas resistant to dopamine agonist therapy or recurrent Cushing's disease during a visit in the clinic office and ask if these subjects would be interested in participating in this study. If the subjects express interest, they will be given the consent form to review. They will be encouraged to review it with family, friends, and/or other physicians. The PI, co-investigators, or research nurse will be available for any questions the subjects might have. If the subjects are still interested, they will be asked to sign and return the consent form to the office and a study visit will be scheduled.

The PI, co-investigator, or member of study staff may also attempt to contact current patients by phone to assess interest in participating in the study. The purpose and overall structure of the study will be discussed with the possible participant. They will be reminded that the study is strictly voluntary and that their involvement or disinterest in the study will not affect their ongoing care. If the patient is interested they will be mailed a consent to review and will be asked to call the center to schedule an appointment to further discuss the study if they decide they are interested.

Each participant will undergo 8 visits of the course of the study. Each participant will have a baseline visit where a medical history will be taken, a physical, visual field test, electrocardiogram (ECG), echocardiogram (ECHO), and blood draw will be performed. At this point lapatinib therapy will begin and the patients will be asked to take the drug daily for the next six months. Patients will take Lapatinib 1250 mg daily (orally), which is the standardized dose used to treat breast cancer patients. Visit 2 will be 1 month after the participant has started lapatinib. At visit 2 all participants will receive a physical exam, a history will be taken, an ECG will be performed, and a blood draw will occur. Visit 3 will be 2 months after starting lapatinib. A physical exam and history will be performed along with an ECG and echocardiogram and blood draw. Visit 4 will be 3 months after starting lapatinib. A physical, history, blood draw, ECG, visual field test, and a magnetic resonance imaging (MRI) of the pituitary will be performed. Visit 5 will occur 4 months after starting lapatinib. A physical exam and history along with a blood draw and ECG and echocardiogram will occur. Visit 6 will be 5 months after starting lapatinib. A physical exam, history, ECG, and a blood draw will occur. Visit 7 will occur 6 months after the start of lapatinib. A physical exam, history, blood draw, visual field test, ECG, echocardiogram and MRI of the pituitary will occur. At this point lapatinib will be discontinued. Visit 8 will occur 1 month after visit 7 and a physical exam, history, blood draw, and ECG and and echocardiogram will occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nonfunctioning adenomas who have undergone at least one prior surgical resection and have demonstrated recurrence on MRI
* Patients with prolactinomas who are resistant to dopamine agonist therapy
* Patients with malignant pituitary tumors
* Patients with visual field deficits and/or compression of the optic chiasm must be stable for at least 6 months

Exclusion Criteria:

* Patients with compromised visual fields and/or compression of the optic chiasm on MRI that has not been stable for last 6 months.
* Patients that have reduced left ventricular ejection fraction less than 50%
* Patients with moderate to severe hepatic impairment
* Patients that are pregnant or lactating
* Patients under the age of 18
* Active hepatitis
* Known previous HIV Positive
* Concurrent cancers
* Life expectancy less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Odelia Cooper, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Dong W, Shi W, Liu Y, Li J, Zhang Y, Dong G, Dong X, Gao H. CHST7 Methylation Status Related to the Proliferation and Differentiation of Pituitary Adenomas. Cells. 2022 Aug 4;11(15):2400. doi: 10.3390/cells11152400. PMID 35954244
- [Derived] Cooper O, Bonert VS, Rudnick J, Pressman BD, Lo J, Salvatori R, Yuen KCJ, Fleseriu M, Melmed S. EGFR/ErbB2-Targeting Lapatinib Therapy for Aggressive Prolactinomas. J Clin Endocrinol Metab. 2021 Jan 23;106(2):e917-e925. doi: 10.1210/clinem/dgaa805. PMID 33150390

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib: All participants will be asked to take Lapatinib 1250 mg po daily for a total of six months during the research study.
  Lapatinib: All participants will be asked to take Lapatinib daily for six months during the research study.
Period: Overall Study
Arm/Group | Lapatinib
Started | 9
Completed | 6
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Prolactin [Mean (Standard Deviation); unit: ng/ml] | 2367 (4617)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Volume
Description: Tumor volume will be assessed on MRI at 6 months on therapy and compared to baseline MRI.
Time Frame: baseline and at 6 months
Population: Note: 1 subject was withdrawn after 6 weeks of lapatinib therapy and therefore not included in analysis. A 2nd subject was not included in this analysis as the drug was given on compassionate basis to prevent recurrence of her tumor. She had a negative baseline MRI and maintained a negative MRI at study end.
Measure: Median (Full Range); unit: Percent volume
Arm/Group | Lapatinib
Number analyzed (Participants) | 7
Percent volume | 10 [-41.4 to 318]

2. Primary Outcome: Number of Participants With 50% Reduction in Prolactin Levels
Description: 50% reduction in prolactin level measured monthly on 6 months therapy compared to baseline level.
Time Frame: every month, up to 6 months
Population: There were 6 prolactinomas and 3 nonfunctioning tumors in this trial. Prolactin results are only reported for the prolactinomas.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 6
Participants | 1

3. Secondary Outcome: % Change in Prolactin From Baseline to Study End
Description: Percent prolactin change from start of lapatinib to end of study participant participation
Time Frame: Baseline and at 6 months
Population: Prolactin results only reported on the 6 prolactinomas in the trial and not for the nonfunctioning tumors.
Measure: Median (Full Range); unit: percent change in prolactin
Arm/Group | Lapatinib
Number analyzed (Participants) | 6
percent change in prolactin | -7.0 [-78.5 to 103.0]

4. Secondary Outcome: ErbB Receptor Expression
Description: Mean percent positive expression of EGFR and ErbB2 will be tested on pathologic tumor specimens from subjects treated with lapatinib
Time Frame: at 6 months
Population: Of the subjects who participated in the trial, only 3 had available tumor tissue to immunostain. Therefore, results could not be reported on the other subjects.
Measure: Mean (Standard Deviation); unit: percent positive expression
Arm/Group | Lapatinib
Number analyzed (Participants) | 3
percent positive expression | 0 (0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 6 months
Description: Prior to initiating therapy, patients were assessed with monthly echocardiogram,ECG, physical examinations, chemistry and hematology panels. Adverse events were graded by the NCI-CTC. Subjects with toxicity equal to Grade 3 on the NCI-CTC will have their dose held and resumed at a fifty percent dose reduction when the toxicity has resolved. Those subjects with toxicity equal to Grade 4 were discontinued on the study drug.
Arm/Group | Lapatinib
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (N=9)
Transaminitis (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (N=9)
Rash (Skin and subcutaneous tissue disorders) | 5 — Acneiform rash noted in 5 subjects
Diarrhea (Gastrointestinal disorders) | 2
Bradycardia (Cardiac disorders) | 3
Transaminitis (Hepatobiliary disorders) | 2

LIMITATIONS AND CAVEATS:
For one of the secondary outcomes, the ErbB receptor expression, only 3 subjects had tumor specimens available to immunostain. Therefore, only results on 3 subjects were reported for this outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT00939523/Prot_SAP_000.pdf